CLINICAL TRIAL: NCT00065338
Title: Nutritional Restriction and Activity Thermogenesis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: James A. Levine, M.D., Ph.D., Consultant, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DK63226 (completed); R01DK063226 (NIH)
Record Dates: First submitted 2003-07-21; First posted 2003-07-23 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Obesity
Keywords: Physical activity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise; Behavior Therapy

INTERVENTIONS:
Behavioral: Exercise and behavior modification — Participants will undergo 1000 kcal/day caloric restriction (relative to experimentally determined weight-maintenance caloric needs) for 8 weeks during one phase of study. Additional 11 week period consists of 8 weeks of caloric restriction with an additional daily walking program.

SUMMARY:
These studies will provide us with enormous insight regarding how obese patients adapt energetically during negative energy balance. We will gain fundamental information regarding the metabolic implications of combining food restriction with a walking program compatible to that advocated by statutory agencies. These studies will lead to improved understanding of the energetic adaptation that occurs during negative energy balance and how best to treat patients with obesity.

ELIGIBILITY:
Ninety sedentary subjects, aged 25-55, who live <10 miles from Rochester will be recruited. This age range has been selected to enable us to study individuals at the peak age-range of obesity and over-weight prevalence and to avoid issues of menopause. Subjects will not be eligible for consideration if they take two or more bouts of exercise/week or participate in sports for more than 2 hours/week. Subjects with predicted weight maintenance energy requirements of <2000 kcal/day will have been excluded at screening. This is because when we come to underfeeding by 1000 kcal/day, we want to avoid feeding any volunteer <1000 kcal/day, for safety & compliance reasons.

(A) LEAN: 30 (15F,15M) lean subjects; BMI <25 kg/m2. Each lean subject will be individually matched for height (+3cm) and age (+3 years) to an obese subject so as to establish comparable groupings for body size. Subjects will have been weight-stable for six months (B) OBESE: 30 (15F,15M) obese subjects; BMI 30-35 kg/m2. Subjects will have been weight-stable for six months (C) POST-OBESE: 30 (15F,15M) patients will have had a previous BMI >30 kg/m2 and a weight loss sufficient to achieve a BMI of <26 kg/m2 maintained for at least 2 months (with weight fluctuation during this period of <1 kg) (94). We will attempt to match these subjects to the obese subjects as described above.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2003-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Non Exercise Activity Thermogenesis | Weeks 2 and 11, each period

SECONDARY OUTCOMES:
Body weight | Daily
Body Composition | Weeks 2 and 11, each period

CONTACTS AND LOCATIONS:
Overall Officials: James A Levine, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Levine JA, Lanningham-Foster LM, McCrady SK, Krizan AC, Olson LR, Kane PH, Jensen MD, Clark MM. Interindividual variation in posture allocation: possible role in human obesity. Science. 2005 Jan 28;307(5709):584-6. doi: 10.1126/science.1106561. PMID 15681386